CLINICAL TRIAL: NCT04696003
Title: Treatment of Classic Mid-trimester Preterm Premature Rupture of Membranes (PPROM) With Oligo/Anhydramnion Between 22/0-26/0 Week of Gestation by Means of Continuous Amnioinfusion: a Multicenter Prospectiv Randomized Trial
Brief Title: Treatment of Classic Mid-trimester PPROM by Means of Continuous Amnioinfusion
Acronym: AmnionFlush
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Michael Tchirikov MD, PhD, Univ.-Prof. Dr. med., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-185
Record Dates: First submitted 2020-12-21; First posted 2021-01-06 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Bronchopulmonary Dysplasia; Necrotizing Enterocolitis; Intracranial Hemorrhages
Keywords: PPROM, Amnion Flush Solution, outcome, amnioinfusion
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Enterocolitis, Necrotizing; Intracranial Hemorrhages; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Intervention Model Description: randomized multicenter controlled trial; two-arm parallel design.
Who Masked: Outcomes Assessor
Masking Description: The neonatal outcome will be evaluated one year after the delivery by the stuff of the University Center of the Clinical Studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The patients with classic PPROM between 22/0-26/0 weeks' gestation with oligo/anhydramnion with standard conservative treatment (7 days Amoxicillin/Clarithromycin therapy or 7 days Amoxicillin and once Azithromycin 1 g per os, and corticosteroids like Celestan®, Essex Pharma, Munich, Germany) as RDS prophylaxis will represent the control group (DGGG Guideline AWMF 015-025, February 2019, Version 1.0). The diagnosis of the PPROM must be not early than 20/0 weeks' gestation.
- Amnion Flush group (continuous amnioinfusion) (Active Comparator): In the "Amnion Flush" group additionally to the standard treatment the amniotic cavity will be punctured with a 18 gauge needle under ultrasound control. The intra-amniotic catheter (0.65 mm Diameter, CE 0481, PakuMed GmbH, Essen, Germany) will be placed under local anesthesia with Xylocaine 1% 10 ml. Amnion Flush Solution (CE 0483, Serumwerk AG Bernburg, Germany) will be carried out with an infusion rate of 100 ml/h (2400 ml/d) under periodic ultrasound using the standard i.v. pump. The deepest pool of amniotic ﬂuid should be stabilized by about 4 cm. The ultrasound control will be performed daily. Induction of the labour or c-section at 34/0 week of gestation or earlier if indicated.
  Interventions: Combination Product: Continuous amnioinfusion with Amnion Flush Solution through the intraamniotic catheter

INTERVENTIONS:
Combination Product: Continuous amnioinfusion with Amnion Flush Solution through the intraamniotic catheter — The amniotic cavity will be punctured with a 18 gauge needle under ultrasound control. The intraamniotic catheter (0.65 mm Diameter, CE 0481, PakuMed GmbH, Essen, Germany) will be placed under local anesthesia with Xylocaine 1% 10 ml. and the amnioinfusion (about 100 ml/h, 2400 ml/day) with artificial amniotic fluid (Amnion Flush Solution, CE 0483, Serumwerk AG Bernburg, Germany) will be carried out with an infusion rate of 100 ml/h under periodic ultrasound using the standard i.v. pump.
  Arms: Amnion Flush group (continuous amnioinfusion)

SUMMARY:
Objective: Mid-trimester preterm premature rupture of membranes (PPROM), defined as rupture of fetal mem-branes prior to 28 weeks' gestation (WG), complicates approximately 0.4-0.7% of all pregnancies and associated with very high neonatal mortality and morbidity. Antibiotics have limited success to prevent bacteremia, chorioamnionitis and fetal inflammation because of reduced placental transport. The repetitive amnioinfusion doesn't work because of immediately fluid lost after the intervention). The continuous amnioinfusion with Amnion Flush Solution through the perinatal port system in patients with classic PPROM prolonged the PPROM-to-delivery interval to 49 days in average by flush out of bacteria and inflammatory components from the amniotic cavity.

Aim: This multicenter trial tests the effect of continuous amnioinfusion on the neonatal survival without major morbidities, like severe bronchopulmonary dysplasia, intraventricular hemorrhage, cystic periventricular leukomalacia and necrotizing enterocolitis.

Design: randomized multicenter controlled trial; two-arm parallel design. Control group: 34 PPROM patients between 22/0 (20/0) -26/0 WG treating with antibiotics and corticosteroids in according to DGGG guide-lines. In interventional group (n=34) the standard PPROM therapy will be complemented by "Amnion -Flush" method with the amnioinfusion of artificial amniotic fluid (Amnion Flush Solution, Serumwerk AG, Germany, 2400 ml/d).

Subjects: Patients with classic PPROM between 22/0-26/0 WG. Expected outcome:The investigators expect significant reduction of neonatal mortality and morbidity in the "Amnion-Flush" group.

DETAILED DESCRIPTION:
Objective:

Mid-trimester preterm premature rupture of membranes (PPROM), defined as rupture of fetal mem-branes prior to 28 weeks' gestation (WG), complicates approximately 0.4-0.7% of all pregnancies and associated with very high neonatal mortality and morbidity. Antibiotics have limited success to prevent bacteremia, chorioamnionitis and fetal inflammation because of reduced placental transport. The repetitive amnioinfusion doesn't work because of immediately fluid lost after the intervention). The continuous amnioinfusion with Amnion Flush Solution through the perinatal port system in patients with classic PPROM prolonged the PPROM-to-delivery interval to 49 days in average by flush out of bacteria and inflammatory components from the amniotic cavity.

Aim: This multicenter trial tests the effect of continuous amnioinfusion on the neonatal survival without major morbidities, like severe bronchopulmonary dysplasia, intraventricular hemorrhage, cystic periventricular leukomalacia and necrotizing enterocolitis.

Design: randomized multicenter controlled trial; two-arm parallel design.

Control group:

34 PPROM patients between 22/0 (20/0) -26/0 WG treating with antibiotics and corticosteroids in according to DGGG guide-lines (7 days Amoxicillin/Clarithromycin therapy or 7 days Amoxicillin and once Azithromycin 1 g and corticosteroids' RDS prophylaxis).

Experimental group:

34 PPROM patients between 22/0 (20/0) -26/0 WG, continuous amnioinfusion (100 ml/h) in pregnant women with classic PPROM with oligo-/anhydramnion between 22/0- 26/0 weeks' gestation and systemic antibiotic therapy (7 days Amoxicil-lin/Clarythromycin or 7 days Amoxicillin and once Azithromycin 1 g) and corticosteroids' RDS prophylaxis.

Duration of intervention: Maximum till 34/0 weeks of gestation, or preterm delivery if indicated.

Follow-up per patient: 12 months post-partum. Subjects: Patients with classic PPROM between 22/0 (20/0) -26/0 WG. Primary efficacy endpoint: survival without major morbidity (severe bron-chopulmonary dysplasia (BPD), and/or grades 3 and 4 intraventricular hemor-rhage (IVH 3-4), and/or cystic periventricular leukomalacia (cPVL), and/or necrotizing enterocolitis (NEC)) since randomization (event time).

Expected outcome: The envestigators expect significant reduction of neonatal mortality and morbidity in the "Amnion-Flush" group.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy (from 22/0 to 26/0 weeks of gestation)
* Evidence of PPROM from clinical and instrumental investigations
* Oligo/anhydramnion (< 2 cm deepest amniotic fluid pocket)

Exclusion Criteria:

* fetal death
* placental abnormalities
* labor
* evidence of major structural or chromosomal abnormalities
* signs of chorioamnionitis (maternal fever > 38° C and one or more of the following criteria: uterine tenderness, malodorous vag-inal discharge, maternal leukocytosis > 15000 cells/mm3, maternal tachycardia > 100 beats/min, and fetal heart rate > 160 bpm).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with bronchopulmonary dysplasia | through study completion, an average of 1 year
  Number of Participants with severe bronchopulmonary dysplasia (BPD)
Number of Participants with intraventricular hemorrhage | through study completion, an average of 1 year
  Number of Participants with intraventricular hemorrhage (IVH 3-4)
Number of Participants with necrotizing enterocolitis | through study completion, an average of 1 year
  Number of Participants with necrotizing enterocolitis (NEC)

SECONDARY OUTCOMES:
Duration of PPROM to delivery interval | up to 15 weeks
  Duration of PPROM to delivbery interval (days)
Gesatational age at delivery | 34 weeks
  gestational age at delivery
Rate of Newborns with FIRS | 1 week
  Rate of Newborns with FIRS (fetal inflammatory response syndrome) (binary)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tchirikov, MD, Ph.D., Study Director — University Clinic of Obstetrics and Prenatal Medicine
Locations (1):
- Martin Luther University, Clinic of Obstetrics and Prenatal Medicine, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tchirikov M, Zhumadilov Z, Winarno AS, Haase R, Buchmann J. Treatment of Preterm Premature Rupture of Membranes with Oligo-/Anhydramnion Colonized by Multiresistant Bacteria with Continuous Amnioinfusion and Antibiotic Administrations through a Subcutaneously Implanted Intrauterine Port System: A Case Report. Fetal Diagn Ther. 2017;42(1):71-76. doi: 10.1159/000438483. Epub 2015 Oct 9. PMID 26447923
- [Background] Tchirikov M, Bapayeva G, Zhumadilov ZSh, Dridi Y, Harnisch R, Herrmann A. Treatment of PPROM with anhydramnion in humans: first experience with different amniotic fluid substitutes for continuous amnioinfusion through a subcutaneously implanted port system. J Perinat Med. 2013 Nov;41(6):657-63. doi: 10.1515/jpm-2012-0296. PMID 23774012
- [Result] Tchirikov M, Schlabritz-Loutsevitch N, Maher J, Buchmann J, Naberezhnev Y, Winarno AS, Seliger G. Mid-trimester preterm premature rupture of membranes (PPROM): etiology, diagnosis, classification, international recommendations of treatment options and outcome. J Perinat Med. 2018 Jul 26;46(5):465-488. doi: 10.1515/jpm-2017-0027. PMID 28710882
- [Derived] Tchirikov M, Haiduk C, Tchirikov M, Riemer M, Bergner M, Li W, Henschen S, Entezami M, Wienke A, Seliger G. Treatment of Classic Mid-Trimester Preterm Premature Rupture of Membranes (PPROM) with Oligo/Anhydramnion between 22 and 26 Weeks of Gestation by Means of Continuous Amnioinfusion: Protocol of a Randomized Multicentric Prospective Controlled TRIAL and Review of the Literature. Life (Basel). 2022 Aug 30;12(9):1351. doi: 10.3390/life12091351. PMID 36143388